CLINICAL TRIAL: NCT01293734
Title: Research on Traditional Chinese Medicine (TCM) Clinical Treatment of the Acute Episode of Bronchial Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Liaoning University of Traditional Chinese Medicine (Other)
Collaborators: Shenyang Huanggu District Central Hospital (Unknown); Benxi City hospital of Chinese medicine (Other); Anshan Central Hospital (Other)
Responsible Party: Zhenwu Guo, No.2 Affiliated Hospital of Liaoning University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sygzwu
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-01

CONDITIONS: Bronchial Asthma
Keywords: bronchial asthma; cold type; heat type; Asthenia type; TCM syndrome; symptoms; physical signs
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- cold type (Experimental): To comply with the diagnostic standard of bronchial asthma in western medicine and TCM syndrome in cold type
  Interventions: Other: warming lung and relieving asthmatic granule and Securing origin and warming lung emplastrum
- heat type (Experimental): To comply with the diagnostic standard of bronchial asthma in western medicine and TCM syndrome in heat type.
  Interventions: Other: clearing lung and relieving asthmatic granule and securing origin and clearing lung emplastrum
- Asthenia type (Experimental): To comply with the diagnostic standard of bronchial asthma in western medicine and TCM syndrome in Asthenia type.
  Interventions: Other: securing origin and relieving asthmatic granule and securing origin and nourishing lung emplastrum
- Western medicine control group (Active Comparator)
  Interventions: Drug: Theophylline Sustained-release Tablets and budesonide suspension

INTERVENTIONS:
Other: warming lung and relieving asthmatic granule and Securing origin and warming lung emplastrum — warming lung and relieving asthmatic granule:once 1 bag, 3 times a day. Securing origin and warming lung emplastrum: paste on acupuncture point and take the emplastrum down after 3 hours, once a day
  Arms: cold type
Other: clearing lung and relieving asthmatic granule and securing origin and clearing lung emplastrum — clearing lung and relieving asthmatic granule: once 1 bag, 3 times a day. securing origin and clearing lung emplastrum: paste on acupuncture point and take the emplastrum down after 3 hours, once a day
  Arms: heat type
Other: securing origin and relieving asthmatic granule and securing origin and nourishing lung emplastrum — securing origin and relieving asthmatic granule: once 1 bag, 3 times a day. securing origin and nourishing lung emplastrum: paste on acupuncture point and take the emplastrum down after 3 hours, once a day
  Arms: Asthenia type
Drug: Theophylline Sustained-release Tablets and budesonide suspension — Theophylline Sustained-release Tablets 0.2g a time, twice a day. budesonide suspension for inhalation 100ug, twice a day
  Arms: Western medicine control group

SUMMARY:
Bronchial asthma is a common disease and frequently encountered disease of respiratory apparatus. It has very complex mechanism and multiple inducing factors. This study will focus on a new Chinese therapy on Bronchial asthma, analyzing the treatment mechanism of internal and external use, based on Traditional Chinese Medicine (TCM) theory and clinical practice. The study will also investigate the efficacy of the Chinese drugs and treatments on Bronchial asthma, and provide an effective therapy for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65 years old;
* Patients with mild-to-moderate bronchial asthma on attacking stage;
* Without cardiopulmonary or other complications;
* To comply with the diagnostic standard of bronchial asthma in western medicine and TCM syndrome differentiation;
* Informed consent form is required to be signed.

Exclusion Criteria:

* Older than 65 years or younger than 18 years old;
* Pregnant woman or suckling period woman;
* Patients combine serious primary disease in liver, renal, cardiovascular and cerebrovascular, hemopoietic system diseases,or psychosis.
* Severe levels of disease is between severe and critical extent. Combine Pulmonary Heart Disease or respiratory failure;
* Irritable the physique, or allergic to the given composition of drugs in this research;
* Patients who are in the process of other clinical research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2008-12; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
primary Symptom | 30 days
  Symptom: wheezing, cough, choking
physical sign | 30 days
  physical sign: wheezing sound
assistant examination | 30 days
  Pulmonary function: mend matters of FEV1, PEF, FEV1/FVC

SECONDARY OUTCOMES:
Secondary Symptom | 30 days
  Symptom: expectoration, fever, Aversion to wind and cold
physical sign | 30 days
  physical sign: tongue appearance and Pulse condition